CLINICAL TRIAL: NCT05361785
Title: Fecal Microbiota Transplantation for Irritable Bowel Syndrome Associated Food Intolerance
Acronym: FinFMT-IBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Turku University Hospital (Other Government); University of Helsinki (Other); Paijat-Hame Hospital District (Other)
Responsible Party: Principal Investigator, Perttu Arkkila, Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1480/2021
Record Dates: First submitted 2022-04-30; First posted 2022-05-05 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Irritable Bowel Syndrome; Fecal Microbiota Transplantation
Keywords: FMT; IBS; FODMAP
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: RCT, randomaization 2/3 FMT, 1/3 placebo
Who Masked: Investigator
Masking Description: Coputer based randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT form healthy donor (Active Comparator): FMT from healthy donor
  Interventions: Biological: FMT
- FMT plasebo (Placebo Comparator): FMT plasebo
  Interventions: Biological: FMT

INTERVENTIONS:
Biological: FMT — FMT from healthy donor or placebo

SUMMARY:
Previous studies have shown that stool transplantation (FMT) have positive effect in symptoms for some patients with irritable bowel syndrome (IBS). Studies have shown that it is possible by FMT to reverse the microbiome of the recipient's intestine in the direction of the microbiome of the donor. The effect on eating habits for engraftment of microbiome by FMT is unknown.

The purpose of this study is to investigate whether FMT relieves FODMAP diet extension without worsening intestinal symptoms in IBS patients.

DETAILED DESCRIPTION:
This is a plasebo controlled study in which we study the effect and safety of FMT in patients who have IBS and have used FODMAP diet. FMT is assessed by colonoscopy route and therafter the patietns receive twice FMT enema from healthy donor or plasebo..

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18-75 years, knowledge of the Finnish language
* IBS patients have been diagnosed with the Rome IV- criteria, all IBS-subtypes will be accepted to the trial
* The patient must consume low FODMAP diet to control IBS symptoms
* Patient must sign the informed consent

Exclusion Criteria:

* Diagnosed allergies to food components in the study dietary protocol
* Pregnancy and breastfeeding
* Antibiotic treatment less than three months prior enrolment
* Faecal incontinence, i.e., inability to retain enema
* Abuse of drugs, alcohol or medications
* Other diagnosis besides IBS causing GI symptoms, these include IBD, microscopic colitis, coeliac disease and bile acid diarrhoea.
* Severe psychiatric or neurologic condition decreasing patient's compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The effect of FMT for tolerance of FODMAPs in the IBS patients' diet | FMT and IBS
  With this study we aim to investigate if FMT treatment promotes inclusion and tolerance of FODMAPs in the IBS patients' diet.

SECONDARY OUTCOMES:
Microbial components explaining the successful broadening of FODMAP diet in IBS patients. | Microbiome and FODMAP
  We aim to investigate what are the microbial components explaining the successful broadening of their diet and identify microbial taxa engrafted from the donor explaining the dietary modifications.
GI symptoms and bacterial fermentaiton status in IBS | Bacterial fermentation status and IBS
  Aim to investigate the gastrointestinal symptom change and see how changes in bacterial fermentation status (detected with hydrogen breath test) modulates the patients' symptoms and if this is related to the FMT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Perttu Arkkila, Professor, Principal Investigator — Head physician; Perttu Lahtinen, Md., Study Chair — Head physician
Locations (1):
- Helsinki University Hospital, Helsinki, Helsinki and Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Yes
Pseudoanonymous data is available to other reserchers
Supporting Information: Study Protocol, CSR
Time Frame: 31 July 2025 for one yrear.
Access Criteria: Scientific work